CLINICAL TRIAL: NCT03512600
Title: Study of the Effects of the Consumption of Different Products Cocoa Derivatives at the Risk of Crystallization of Uric Acid in Urine of Volunteers.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Devicare S.L. (Industry)
Collaborators: Universidad de las Islas Baleares (Unknown)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: IB 3475/17
Record Dates: First submitted 2018-03-23; First posted 2018-05-01 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Lithiasis, Urinary
Keywords: lithiasis; uric acid; crystallization
MeSH Terms: conditions — Urolithiasis; Lithiasis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group (Experimental): All patients will follow four different dietary interventions (with or without cacao) for 1 day prior to the taking of a urine sample.
  After the sample is taken the patient will follow a washout period of 6 days before following a different diet and this process will be repeated for each patient until they have followed the four diets.
  .
  Interventions: Dietary Supplement: Intervention 0; Dietary Supplement: Intervention 1; Dietary Supplement: Intervention 2; Dietary Supplement: Intervention 3

INTERVENTIONS:
Dietary Supplement: Intervention 0 — Without nutritional intervention, it will consist of normal food intake without food derived from cocoa or coffee for a period of 1 day in the group of 20 patients during meals. ( That day the patient can not consume cocoa derivates nor coffe or coffe derivates).
  Other Names: Study group
Dietary Supplement: Intervention 1 — The nutritional intervention will consist of the intake of 40 g daily a base of food derived from cocoa that will be provided to the paient (Food based on soluble cocoa) during one 1 day period in the group of 20 patients during meals.
  That day the patient can not consume cocoa derivates nor coffe or coffe derivates exept the one provided.
  Other Names: Study group
Dietary Supplement: Intervention 2 — The nutritional intervention will consist of the intake of 40 g daily a base of food derived from cacao (Food based on black chocolate) during a period of 1 day in the group of 20 patients during meals.
  That day the patient can not consume cocoa derivates nor coffe or coffe derivates exept the one provided.
  Other Names: Study Group
Dietary Supplement: Intervention 3 — The nutritional intervention will consist of the intake of 40 g daily a base of food derived from cocoa (Food based on chocolate with milk) for a period of 1 day in the group of 20 patients during meals.
  That day the patient can not consume cocoa derivates nor coffe or coffe derivates exept the one provided.
  Other Names: Study group

SUMMARY:
The present study aims to assess the effectiveness of theobromine, -product present in high proportion in the cacao-, to prevent the development of uric acid kidney stones.

DETAILED DESCRIPTION:
Renal lithiasis is a pathology that affects a high percentage of the population, and although it has been known for a long time, advances carried out in the treatment are limited to the surgical aspects, while the causes responsible for the formation of kidney calculus are not corrected, which leads to a high recurrence.

The "healing" of renal lithiasis inevitably goes through the elimination of the alterations related to the genesis of kidney calculus. It the case of uric acid lithiasis the most important are having urinary pH less than 5.5 and an elevated uricosuria, which can be corrected relatively easy by undergoing changes in dietary habits, and with pharmacological treatment with citrate -which produces and increase in pH- or with inhibitors of the xantino-oxidase as allopurinol. However, among the prophylactic treatments available for ural acid lithiasis, so far it does not exist one for urinary acid crystallization inhibition.

Recently, the effects of theobromine as an inhibitor of the crystallization of uric acid have been described, but only in vitro. The present study aims to assess the effectiveness of theobromine, -product present in high proportion in the cacao-, to prevent the development of uric acid kidney stones.

The study is a unicentric, low intervention, non-randomized, prospective study to assess the effects of the consumption of different cocoa derivate products, in the risk of crystallization of uric acid in the urine. Participants in the study are healthy volunteers and will it will be carried out with 20 individuals who will be recruited in the Research Laboratory in Renal Lithiasis of the Baleares Isles University.

Patients will take a urine test previously to undergo 4 dietary interventions, with their subsequent urine measurements. Patients will choose one diet to follow for 1 day, and will be provided with the corresponding cocoa derivate for the diet (soluble cocoa, black chocolate, chocolate with milk). The day after the diet they will take a fast-picking of urine accumulated during the night of which they followed the controlled diet (12 h nocturne sample), then follow a 6 day washout period, and select another diet to follow and repeat until they have gone through the 4 diets and measurements.

ELIGIBILITY:
Inclusion Criteria:

* Compliance in participating and collaborating in the study

Exclusion Criteria:

* Cocoa / chocolate allergy or theobromine
* Pregnancy, nursing period (women)
* pharmacological treatment
* chronic diseases (diabetes, kidney failure, heart failure, hyperuricemia, ...)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-09-04 (Actual); Primary Completion 2017-10-06 (Actual); Study Completion 2017-10-06 (Actual)

PRIMARY OUTCOMES:
Ability to inhibit the crystallization of uric acid in urine collected. | 12 hours
  Ability to inhibit the crystallization of uric acid in urine collected.

SECONDARY OUTCOMES:
Concentration of theobromine in urine. | 12 hours
  Concentration of theobromine in urine.

CONTACTS AND LOCATIONS:
Overall Officials: Fèlix Grases Freixedas, Principal Investigator — Universidad de las Islas Baleares
Locations (1):
- Universitat de les Illes Balears, IUNICS, Palma de Mallorca, Balearic Islands, Spain

IPD SHARING:
Plan to Share IPD: No